CLINICAL TRIAL: NCT04217889
Title: Study of the Adherence to Chest Physiotherapy in Patients With Cystic Fibrosis (CF) at the Adult CF Center in Lyon
Brief Title: Cystic Fibrosis Adherence Study
Acronym: KINOBS
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL19_0410
Record Dates: First submitted 2020-01-02; First posted 2020-01-06 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis; Adherence to chest physiotherapy
MeSH Terms: conditions — Cystic Fibrosis | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Adherent patient: This group is composed of adherent patients to the chest physiotherapy based on the number of chest physiotherapy session per week.
  Interventions: Other: Questionnaire
- Not-adherent patient: This group is composed of not-adherent patients to the chest physiotherapy based on the number of chest physiotherapy session per week.
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Short questionnaire that can be completed during the usual consultation.

SUMMARY:
This study aims to assess the role of some factors which can influence the chest physiotherapy adherence in adult with cystic fibrosis.

At first, we are going to try to consider the adherence of chest physiotherapy. Then, after dividing the patients into two groups - adherent or not adherent - we will attempt to identify the factors which can influence this adherence.

It consists in a short questionnaire that the patient will fill during usual visits.

The hypothesis is that the following factors can play a role in adherence of chest physiotherapy:

* Age
* Age of diagnostic
* Sex
* Fev1
* Number of antibiotic course
* Anxiety/depression
* Work time
* Socio-professional category
* Individual situation
* Physiotherapy with liberal physiotherapist and transport time
* Sport practice
* Family support
* Feeling of work time burden
* Feeling of physiotherapy efficiency
* Feeling of physiotherapy burden

ELIGIBILITY:
Inclusion Criteria:

* respiratory symptoms
* subnormal respiratory function (FEV1 < 80%)
* without lung transplant

Exclusion Criteria:

* lung transplantation approach

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cohort of adult patients with cystic fibrosis and follow-up at the Lyon Reference Center.
Sampling Method: Non-Probability Sample
Enrollment: 197 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-06-02 (Actual); Study Completion 2020-06-02 (Actual)

PRIMARY OUTCOMES:
Quantity of chest physiotherapy | 8 months
  If the quantity of chest physiotherapy alone (do well) or/and with physiotherapist is above or egal at 3 per week, the patient is "adherent" If the quantity of chest physiotherapy is under 3 sessions per week, the patient is "not- adherent" Then we measure the proportion of each group for each secondary factors.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre de Référence de la Mucoviscidose Lyon à l'hôpital Lyon Sud, Pierre-Bénite, France